CLINICAL TRIAL: NCT06429787
Title: Post Marketing Observational Study on Safety of BALFAXAR® vs. KCENTRA for Reversal of Vitamin K Antagonist Induced Anticoagulation in Adults Undergoing Urgent Surgery or Invasive Procedure.
Brief Title: Post Marketing Observational Study on Safety of BALFAXAR vs. KCENTRA for Reversal of Vitamin K Antagonist Induced Anticoagulation in Adults Undergoing Urgent Surgery or Invasive Procedure
Status: Recruiting | Type: Observational
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Other Study IDs: LEX-212
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Vitamin K-Dependent Coagulation Defect; Significant Bleeding Risk
MeSH Terms: conditions — Vitamin K-Dependent Clotting Factors, Combined Deficiency Of, 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BALFAXAR® (500 IU): BALFAXAR will be administered by intravenous (IV) infusion at a rate of 0.12 mL/kg/min (~3 units/kg/min), up to a maximum rate of 8.4 mL/min (~210 units/min). Dosing is individualized based on the patient's baseline International Normalized Ratio (INR) value and body weight
  Interventions: Drug: Balfaxar
- Kcentra® (500 IU): KCENTRA will be administered by intravenous infusion at of 0.12 mL/kg/min (~3 units/kg/min) up to a maximum rate of 8.4 mL/min (~210 units/min). Dosing is individualized based on the patient's baseline International Normalized Ratio (INR) value and body weight.
  Interventions: Drug: Kcentra

INTERVENTIONS:
Drug: Balfaxar — BALFAXAR (prothrombin complex concentrate, human-lans) is a blood coagulation factor replacement product indicated for the urgent reversal of acquired coagulation factor deficiency induced by Vitamin K antagonist (VKA, e.g., warfarin) therapy in adult patients with need for an urgent surgery/invasive procedure
  Groups: BALFAXAR® (500 IU)
Drug: Kcentra — KCENTRA, Prothrombin Complex Concentrate (Human), is a blood coagulation factor replacement product indicated for the urgent reversal of acquired coagulation factor deficiency induced by Vitamin K antagonist (VKA, e.g., warfarin) therapy in adult patients with:
  * acute major bleeding or
  * need for an urgent surgery/invasive procedure
  Groups: Kcentra® (500 IU)

SUMMARY:
Post marketing observational study on safety of BALFAXAR vs. KCENTRA for Reversal of Vitamin K Antagonist Induced Anticoagulation in Adults Undergoing Urgent Surgery or Invasive Procedure

ELIGIBILITY:
Inclusion Criteria:

1. Subjects at least 18 years of age.
2. Subjects on VKA treatment.
3. Received 4F-PCC agent, BALFAXAR or Kcentra, for urgent reversal of within 48 hours prior to urgent surgery or invasive procedure.

Exclusion Criteria:

1. History of TEE within 90 days before receipt of VKA reversal therapy.
2. Subjects treated with VKA reversal therapy and not undergoing urgent invasive procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at least 18 years of age who are currently on Vitamin K Antagonist treatments and received BALFAXAR or Kcentra for urgent reversal of VKA therapy within 48 hours prior to urgent surgery or invasive procedure. Octapharma will not actively enroll any of the 3,574 projected subjects into the study. Subjects meeting the minimum inclusion and exclusion criteria during the course of routine practice will be added to the study on a monthly basis until the sample size required for the analysis is achieved in each group.
Sampling Method: Probability Sample
Enrollment: 3574 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
TEEs within 45 days following VKA reversal treatment | 45 days
  Proportion of subjects diagnosed with TEEs within 45 days following VKA reversal treatment with BALFAXAR compared to proportion of subjects diagnosed with TEEs within the same period following VKA reversal treatment with Kcentra.

SECONDARY OUTCOMES:
TEEs within 7 and 14 days following VKA reversal treatment | 14 days
  Proportion of subjects diagnosed with TEEs within 7 and 14 days following VKA reversal treatment with BALFAXAR compared to proportion of subjects diagnosed with TEEs within the same period following VKA reversal treatment with Kcentra.
Median Time to TEEs | 45 days
  Median time to TEE following administration of BALFAXAR compared to median time to TEE following administration of Kcentra
All Cause Mortality | 45 days
  Proportion of subjects who die from any reason within 7, 14 and 45 days following VKA reversal treatment with BALFAXAR compared to proportion of subjects who die from any reason within the same time period following treatment with Kcentra.
Median Time to All Cause Mortality | 45 days
  Median time to death following administration of BALFAXAR compared to median time to death following administration of Kcentra
Rate of Fatal TEEs | 45 days
  Rate of fatal TEEs following treatment with BALFAXAR compared to rate of fatal TEEs following treatment with Kcentra within 7, 14 and 45 days following VKA reversal treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Octapharma Research Site, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No